CLINICAL TRIAL: NCT02307435
Title: Potency of Allogenic Bone Marrow, Umbilical Cord, Adipose Mesenchymal Stem Cell for Non Union Fracture and Long Bone Defect, Directly and Cryopreserved
Brief Title: Allogenic Mesenchymal Stem Cell for Bone Defect or Non Union Fracture
Acronym: AMSC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ismail Hadisoebroto Dilogo, orthopaedic medical doctor, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISMMSC001
Record Dates: First submitted 2014-10-07; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Non Union Fracture; Metaphyseal Fibrous Defect
Keywords: non union fracture; bone defect; mesenchymal stem cell; cryopreservation
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- implantation group (Experimental): implantation group will receive MSC and HA-CaSo4
  Interventions: Biological: MSC

INTERVENTIONS:
Biological: MSC — subjects are implanted with allogenic mesenchymal stem cells from umbilical cord/ bone marrow/ adipose

SUMMARY:
Mesenchymal stem cell (MSC) is one kind of stem cell which is gained form adult tissue. Although MSC derived from autogenic bone marrow are proven to help regeneration in non union fracture and long bone defect, the aspiration process through iliac crest is invasive and painful.

Therefore, alternative source of MSC which is less invasive is needed. Adipose and umbilical cord is a "waste product" that proven to contain enormous MSC. Furthermore adipose and umbilical cord as an allogenic source is more abundant in number compares to autogenic bone marrow. This enormous source need and adequate preservation technique before applied to the patient. According to that, researchers want to explore the potency of MSC from bone marrow, umbilical cord and adipose as the source of allogenic MSC and the effect of cryopreservation technique to the viability and quality of MSC. We will also compare the effectivity of MSC implantation from bone marrow, umbilical cord and adipose applied to non union fracture and long bone defect.

Samples from bone marrow, umbilical cord and adipose are cultured and the viability of the cells are observed. Some of the cells are implanted directly to the patient with non union fractures and long bone defect while some are cryopreserved in liquid nitrogen -190 degree Celsius in three months. All samples are thawed and the viability of the cells are observed. Patient who are implanted by MSC allogenic will undergo clinical and radiological examination in the third, sixth and twenty second month after implantation.

DETAILED DESCRIPTION:
Research Methods Study Design This study is an experimental one arm study post test only. Estimated Study Time Research estimated time would be 24 months, from May 2014 to May 2016. Sample Gaining Procedure This research is a pilot study. Samples are obtained consecutively from all source population that meet the criteria. The number of samples from each mesenchymal stem cell ( adipose, bone marrow and umbilical cord) source are three. Each samples derived from three different donors that met the inclusion criteria. For the implanation, the subjects are five from each intervention. Yet regarding the limited funding source and time, we will recruit one subject for each kind of MSC.

Subject Criteria Inclusion criteria for MSC donor

Bone marrow donor :

Male/female aged 19-30 year without any comorbiditites (Diabetes mellitus, cardiovascular and any other autoimmune disease), HIV test Hepatitis B test and Hepatitis C test are negaitve, no fungal and bacterial contamination in the bone marrow. Subjects are willing to be aspiratied in the iliac crest in order to get the bone marrow.

Adipose donor :

Adipose tissue are gained from liposuction or open reduction internal fixation procedure. Samples of adipose are free from HIV, Hepatitis B, Hepatitis C and free from fungal and bacterial contamination.

Umbilical cord donor :

Umbilical cord are form elective seccio caecaria from a fullterm mother without any complications and free from HIV, hepatitis B, hepatitis C and no fungal and bacterial contamination.

Recipient inclusion criteria Critical bone defect patients aged 6-55 who are willing to undergo surgical intervention.

Recipient exclusion criteria Patients with pathological fracture caused by malignancy, immunocompromised ( HIV AIDS, Diabetes mellitus, active Hepatitis), in a immunosuppresant therapy ( chemotherapy or steroids).

Drop out criteria Patients are ruled out from this study if he/she stated to do so in the time this research are held or she/he undergoes any other threatment that are not related to this study. Patient who does not show any clinical improvement in three consecutive months is categorized as failed to threat. All drop out and failed to threat patient could get other threatment.

Informed Consent All subjects must fill and sign in the informed consent letters.

Research Protocol Mesenchymal stem cell taking method Bone Marrow taking Patient is lying down in supine position, anesthetized locally. Aseptic and antiseptic are done in the illiac crest location. Aspiration needle is inserted 450 to horizon in illiac crest. Hub is released and a 10 cc syringe that contain heparin is connected to te needle. We aspirated about 50 cc bone marrow from each subject.

Umbilical cord taking Right after the delivering the baby, the umbilical cord are cut and kept in a sterile bowl containing 0.9% NaCl in 40 until the sample is proceed.

Adipose taking Adipose tissue are derived from liposuction or open reduction internal fixation procedure. It is kept in a sterile bowl containing NaCL 0.9% in 40 C. Processing of the sample is done within 8 hours after sample are taken.

Cryopreservation and re activation. All the samples are taken to culture laboratory in integrated service of stem cell medical technology Cipto mangunkusumo hospita.this laboratory is GMP (good manufacturing Product) certified. The samples ate cultured in appropriated medium until it reach confluence and harvested. The cells then undergo caracterisation test by flow cyto meter and viability and numbers are counted. Some of the cells then cryopreserved while some are directly implanted into patient. The cells are cryopreserved for three months and then reactivated. Viability and numbers then are measured. The cells then are implanted to non union patient.

Specimen sterility Sterility tests are done three times to ensure there is no fungal and bacterial contamination.

HA-CaSO4 and MSC For every centimeter of defect, 10 millions cells and 50 pellet HA-CaSO4 are needed. The diluted MSC then mix with the HA-CaSO4 and incubated 5 minutes before implanted.

Intervention Surgical intervention is needed to assemble the fixation device in the long bone. During the surgery, pellet HA-CaSO4 are inserted into the defect. After soft tissue are closed the rest of the serum is injected into the defect area.

Observation and follow up Clinical and radiological follow up is done every 4 weeks. Observation is done for 12 months or untill the bone unites. Every subject will be followed up in the third, sixth, twelfth and twenty forth or until the fixation device is taken off.

Recipient criteria for non union fracture

ELIGIBILITY:
Inclusion criteria for MSC donor

* Bone marrow donor : Male/female aged 19-30 year without any comorbiditites (Diabetes mellitus, cardiovascular and any other autoimmune disease),HIV test Hepatitis B test and Hepatitis C test are negaitve, no fungal and bacterial contamination in the bone marrow. Subjects are willing to be aspiratied in the iliac crest in order to get the bone marrow.
* Adipose donor : Adipose tissue are gained from liposuction or open reduction internal fixation procedure. Samples of adipose are free from HIV, Hepatitis B, Hepatitis C and free from fungal and bacterial contamination.
* Umbilical cord donor : Umbilical cord are form elective seccio caecaria from a fullterm mother without any complications and free from HIV, hepatitis B, hepatitis C and no fungal and bacterial contamination.

exclusion / Drop out criteria

-Patients are ruled out from this study if he/she stated to do so in the time this research are held or she/he undergoes any other threatment that are not related to this study. Patient who does not show any clinical improvement in three consecutive months is categorized as failed to threat. All drop out and failed to threat patient could get other threatment.

inclusion criteria for recipient : -male/female aged 6-55 year old with bone critical defect

exclusion criteria for recipient :

-Patients with pathological fracture caused by malignancy, immunocompromised ( HIV AIDS, Diabetes mellitus, active Hepatitis), in a immunosuppresant therapy ( chemotherapy or steroids).

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
cell viability | 3 months
  percentage of cells that live divided by total cell

SECONDARY OUTCOMES:
lower extremity functional score | 3 months
  lower extremities functional score sheet
disabilities of arm shoulder and hand | 3 months
  disabilities of arm shoulder and hand score

CONTACTS AND LOCATIONS:
Overall Officials: ISMAIL H DILOGO, MD, Principal Investigator — integrated unit of stem cell and medical technology CIPTO MANGUNKUSUMO GENERAL HOSPITAL, FACULTY OF MEDICINE UNIVERSITI OF INDONESIA, INDONESIA; ismail h dilogo, MD, Principal Investigator — Indonesia University
Locations (2):
- Indonesia (2):
  - University of Indonesia, Jakarta Pusat, Jakarta Special Capital Region
  - Faculty of Medicine, University of Indonesia, Propinsi DKI Jakarta, Jakarta Special Capital Region

REFERENCES:
- [Background] Kon E, Muraglia A, Corsi A, Bianco P, Marcacci M, Martin I, Boyde A, Ruspantini I, Chistolini P, Rocca M, Giardino R, Cancedda R, Quarto R. Autologous bone marrow stromal cells loaded onto porous hydroxyapatite ceramic accelerate bone repair in critical-size defects of sheep long bones. J Biomed Mater Res. 2000 Mar 5;49(3):328-37. doi: 10.1002/(sici)1097-4636(20000305)49:33.0.co;2-q. PMID 10602065
- [Background] Hee HT, Ismail HD, Lim CT, Goh JC, Wong HK. Effects of implantation of bone marrow mesenchymal stem cells, disc distraction and combined therapy on reversing degeneration of the intervertebral disc. J Bone Joint Surg Br. 2010 May;92(5):726-36. doi: 10.1302/0301-620X.92B5.23015. PMID 20436013
- [Background] Ye Z, Wang Y, Xie HY, Zheng SS. Immunosuppressive effects of rat mesenchymal stem cells: involvement of CD4+CD25+ regulatory T cells. Hepatobiliary Pancreat Dis Int. 2008 Dec;7(6):608-14. PMID 19073406
- [Background] Bocelli-Tyndall C, Bracci L, Spagnoli G, Braccini A, Bouchenaki M, Ceredig R, Pistoia V, Martin I, Tyndall A. Bone marrow mesenchymal stromal cells (BM-MSCs) from healthy donors and auto-immune disease patients reduce the proliferation of autologous- and allogeneic-stimulated lymphocytes in vitro. Rheumatology (Oxford). 2007 Mar;46(3):403-8. doi: 10.1093/rheumatology/kel267. Epub 2006 Aug 18. PMID 16920750
- [Background] Yanez R, Lamana ML, Garcia-Castro J, Colmenero I, Ramirez M, Bueren JA. Adipose tissue-derived mesenchymal stem cells have in vivo immunosuppressive properties applicable for the control of the graft-versus-host disease. Stem Cells. 2006 Nov;24(11):2582-91. doi: 10.1634/stemcells.2006-0228. Epub 2006 Jul 27. PMID 16873762
- [Background] Tipnis S, Viswanathan C, Majumdar AS. Immunosuppressive properties of human umbilical cord-derived mesenchymal stem cells: role of B7-H1 and IDO. Immunol Cell Biol. 2010 Nov-Dec;88(8):795-806. doi: 10.1038/icb.2010.47. Epub 2010 Apr 13. PMID 20386557
- [Result] Hou ZL, Liu Y, Mao XH, Wei CY, Meng MY, Liu YH, Zhuyun Yang Z, Zhu H, Short M, Bernard C, Xiao ZC. Transplantation of umbilical cord and bone marrow-derived mesenchymal stem cells in a patient with relapsing-remitting multiple sclerosis. Cell Adh Migr. 2013 Sep-Oct;7(5):404-7. doi: 10.4161/cam.26941. Epub 2013 Oct 30. PMID 24192520
- [Result] Brinker MR, O'Connor DP. The incidence of fractures and dislocations referred for orthopaedic services in a capitated population. J Bone Joint Surg Am. 2004 Feb;86(2):290-7. PMID 14960673
- [Result] Liebergall M, Schroeder J, Mosheiff R, Gazit Z, Yoram Z, Rasooly L, Daskal A, Khoury A, Weil Y, Beyth S. Stem cell-based therapy for prevention of delayed fracture union: a randomized and prospective preliminary study. Mol Ther. 2013 Aug;21(8):1631-8. doi: 10.1038/mt.2013.109. Epub 2013 Jun 4. PMID 23732992
- [Result] Sen MK, Miclau T. Autologous iliac crest bone graft: should it still be the gold standard for treating nonunions? Injury. 2007 Mar;38 Suppl 1:S75-80. doi: 10.1016/j.injury.2007.02.012. PMID 17383488
- [Result] Goulet JA, Senunas LE, DeSilva GL, Greenfield ML. Autogenous iliac crest bone graft. Complications and functional assessment. Clin Orthop Relat Res. 1997 Jun;(339):76-81. doi: 10.1097/00003086-199706000-00011. PMID 9186204
- [Result] Mauney JR, Volloch V, Kaplan DL. Role of adult mesenchymal stem cells in bone tissue engineering applications: current status and future prospects. Tissue Eng. 2005 May-Jun;11(5-6):787-802. doi: 10.1089/ten.2005.11.787. PMID 15998219
- [Result] Cavallo C, Cuomo C, Fantini S, Ricci F, Tazzari PL, Lucarelli E, Donati D, Facchini A, Lisignoli G, Fornasari PM, Grigolo B, Moroni L. Comparison of alternative mesenchymal stem cell sources for cell banking and musculoskeletal advanced therapies. J Cell Biochem. 2011 May;112(5):1418-30. doi: 10.1002/jcb.23058. PMID 21321995
- [Result] Jurgens WJ, Oedayrajsingh-Varma MJ, Helder MN, Zandiehdoulabi B, Schouten TE, Kuik DJ, Ritt MJ, van Milligen FJ. Effect of tissue-harvesting site on yield of stem cells derived from adipose tissue: implications for cell-based therapies. Cell Tissue Res. 2008 Jun;332(3):415-26. doi: 10.1007/s00441-007-0555-7. Epub 2008 Apr 1. PMID 18379826
- [Result] Lu Z, Wang G, Dunstan CR, Chen Y, Lu WY, Davies B, Zreiqat H. Activation and promotion of adipose stem cells by tumour necrosis factor-alpha preconditioning for bone regeneration. J Cell Physiol. 2013 Aug;228(8):1737-44. doi: 10.1002/jcp.24330. PMID 23359411
- [Result] Parolini O, Alviano F, Bagnara GP, Bilic G, Buhring HJ, Evangelista M, Hennerbichler S, Liu B, Magatti M, Mao N, Miki T, Marongiu F, Nakajima H, Nikaido T, Portmann-Lanz CB, Sankar V, Soncini M, Stadler G, Surbek D, Takahashi TA, Redl H, Sakuragawa N, Wolbank S, Zeisberger S, Zisch A, Strom SC. Concise review: isolation and characterization of cells from human term placenta: outcome of the first international Workshop on Placenta Derived Stem Cells. Stem Cells. 2008 Feb;26(2):300-11. doi: 10.1634/stemcells.2007-0594. Epub 2007 Nov 1. PMID 17975221
- [Result] Troyer DL, Weiss ML. Wharton's jelly-derived cells are a primitive stromal cell population. Stem Cells. 2008 Mar;26(3):591-9. doi: 10.1634/stemcells.2007-0439. Epub 2007 Dec 6. PMID 18065397
- [Result] Bernardo ME, Emons JA, Karperien M, Nauta AJ, Willemze R, Roelofs H, Romeo S, Marchini A, Rappold GA, Vukicevic S, Locatelli F, Fibbe WE. Human mesenchymal stem cells derived from bone marrow display a better chondrogenic differentiation compared with other sources. Connect Tissue Res. 2007;48(3):132-40. doi: 10.1080/03008200701228464. PMID 17522996
- [Result] Im GI, Shin YW, Lee KB. Do adipose tissue-derived mesenchymal stem cells have the same osteogenic and chondrogenic potential as bone marrow-derived cells? Osteoarthritis Cartilage. 2005 Oct;13(10):845-53. doi: 10.1016/j.joca.2005.05.005. PMID 16129630
- [Result] Jin HJ, Bae YK, Kim M, Kwon SJ, Jeon HB, Choi SJ, Kim SW, Yang YS, Oh W, Chang JW. Comparative analysis of human mesenchymal stem cells from bone marrow, adipose tissue, and umbilical cord blood as sources of cell therapy. Int J Mol Sci. 2013 Sep 3;14(9):17986-8001. doi: 10.3390/ijms140917986. PMID 24005862
- [Result] Kern S, Eichler H, Stoeve J, Kluter H, Bieback K. Comparative analysis of mesenchymal stem cells from bone marrow, umbilical cord blood, or adipose tissue. Stem Cells. 2006 May;24(5):1294-301. doi: 10.1634/stemcells.2005-0342. Epub 2006 Jan 12. PMID 16410387
- [Result] Miao Z, Jin J, Chen L, Zhu J, Huang W, Zhao J, Qian H, Zhang X. Isolation of mesenchymal stem cells from human placenta: comparison with human bone marrow mesenchymal stem cells. Cell Biol Int. 2006 Sep;30(9):681-7. doi: 10.1016/j.cellbi.2006.03.009. Epub 2006 Apr 22. PMID 16870478
- [Result] Hu L, Hu J, Zhao J, Liu J, Ouyang W, Yang C, Gong N, Du L, Khanal A, Chen L. Side-by-side comparison of the biological characteristics of human umbilical cord and adipose tissue-derived mesenchymal stem cells. Biomed Res Int. 2013;2013:438243. doi: 10.1155/2013/438243. Epub 2013 Jul 7. PMID 23936800 (Retraction: PMID 33178822 Biomed Res Int. 2020 Sep 23;2020:3176431)
- [Result] Toupadakis CA, Wong A, Genetos DC, Cheung WK, Borjesson DL, Ferraro GL, Galuppo LD, Leach JK, Owens SD, Yellowley CE. Comparison of the osteogenic potential of equine mesenchymal stem cells from bone marrow, adipose tissue, umbilical cord blood, and umbilical cord tissue. Am J Vet Res. 2010 Oct;71(10):1237-45. doi: 10.2460/ajvr.71.10.1237. PMID 20919913
- [Result] Shafiee A, Seyedjafari E, Soleimani M, Ahmadbeigi N, Dinarvand P, Ghaemi N. A comparison between osteogenic differentiation of human unrestricted somatic stem cells and mesenchymal stem cells from bone marrow and adipose tissue. Biotechnol Lett. 2011 Jun;33(6):1257-64. doi: 10.1007/s10529-011-0541-8. Epub 2011 Feb 2. PMID 21287233
- [Result] Arinzeh TL, Peter SJ, Archambault MP, van den Bos C, Gordon S, Kraus K, Smith A, Kadiyala S. Allogeneic mesenchymal stem cells regenerate bone in a critical-sized canine segmental defect. J Bone Joint Surg Am. 2003 Oct;85(10):1927-35. doi: 10.2106/00004623-200310000-00010. PMID 14563800
- [Result] Bruder SP, Kraus KH, Goldberg VM, Kadiyala S. The effect of implants loaded with autologous mesenchymal stem cells on the healing of canine segmental bone defects. J Bone Joint Surg Am. 1998 Jul;80(7):985-96. doi: 10.2106/00004623-199807000-00007. PMID 9698003
- [Result] Viateau V, Guillemin G, Bousson V, Oudina K, Hannouche D, Sedel L, Logeart-Avramoglou D, Petite H. Long-bone critical-size defects treated with tissue-engineered grafts: a study on sheep. J Orthop Res. 2007 Jun;25(6):741-9. doi: 10.1002/jor.20352. PMID 17318898
- [Result] Schubert T, Lafont S, Beaurin G, Grisay G, Behets C, Gianello P, Dufrane D. Critical size bone defect reconstruction by an autologous 3D osteogenic-like tissue derived from differentiated adipose MSCs. Biomaterials. 2013 Jun;34(18):4428-38. doi: 10.1016/j.biomaterials.2013.02.053. Epub 2013 Mar 16. PMID 23507085
- [Result] Shoji T, Ii M, Mifune Y, Matsumoto T, Kawamoto A, Kwon SM, Kuroda T, Kuroda R, Kurosaka M, Asahara T. Local transplantation of human multipotent adipose-derived stem cells accelerates fracture healing via enhanced osteogenesis and angiogenesis. Lab Invest. 2010 Apr;90(4):637-49. doi: 10.1038/labinvest.2010.39. Epub 2010 Feb 15. PMID 20157290
- [Result] Thirumala S, Goebel WS, Woods EJ. Clinical grade adult stem cell banking. Organogenesis. 2009 Jul;5(3):143-54. doi: 10.4161/org.5.3.9811. PMID 20046678
- [Result] Matsumura K, Hayashi F, Nagashima T, Hyon SH. Long-term cryopreservation of human mesenchymal stem cells using carboxylated poly-l-lysine without the addition of proteins or dimethyl sulfoxide. J Biomater Sci Polym Ed. 2013;24(12):1484-97. doi: 10.1080/09205063.2013.771318. Epub 2013 Feb 22. PMID 23829460
- [Result] Dariolli R, Bassaneze V, Nakamuta JS, Omae SV, Campos LC, Krieger JE. Porcine adipose tissue-derived mesenchymal stem cells retain their proliferative characteristics, senescence, karyotype and plasticity after long-term cryopreservation. PLoS One. 2013 Jul 9;8(7):e67939. doi: 10.1371/journal.pone.0067939. Print 2013. PMID 23874472
- [Result] Angelo PC, Ferreira AC, Fonseca VD, Frade SP, Ferreira CS, Malta FS, Pereira AK, Leite HV, Brum AP, Pardini VC, Gomes KB, Cabral AC. Cryopreservation does not alter karyotype, multipotency, or NANOG/SOX2 gene expression of amniotic fluid mesenchymal stem cells. Genet Mol Res. 2012 Apr 19;11(2):1002-12. doi: 10.4238/2012.April.19.5. PMID 22576926
- [Result] Park M, Seo JJ. Role of HLA in Hematopoietic Stem Cell Transplantation. Bone Marrow Res. 2012;2012:680841. doi: 10.1155/2012/680841. Epub 2012 Oct 2. PMID 23082252
- [Result] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Result] Liu LY, Chai JK, Duan HJ, Hou YS, Yin HN, Yu YH, Hu Q, Hao DF, Feng G, Li T, Du JD. [Comparison of different methods for the isolation of human umbilical cord mesenchymal stem cells]. Zhonghua Yi Xue Za Zhi. 2013 Aug 27;93(32):2592-6. Chinese. PMID 24351605
- [Result] Han ZX, Shi Q, Wang DK, Li D, Lyu M. [Basic biological characteristics of mesenchymal stem cells derived from bone marrow and human umbilical cord]. Zhongguo Shi Yan Xue Ye Xue Za Zhi. 2013 Oct;21(5):1248-55. doi: 10.7534/j.issn.1009-2137.2013.05.033. Chinese. PMID 24156444